CLINICAL TRIAL: NCT00258999
Title: Predictor of Advanced Sub-Clinical Atherosclerosis (PASA) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2005-0342
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2007-12

CONDITIONS: Atherosclerosis
Keywords: Skin Cholesterol; Carotid Plaque; Carotid Intima-Media Thickness
MeSH Terms: conditions — Atherosclerosis

INTERVENTIONS:
Device: Skin Cholesterol Testing

SUMMARY:
The study will evaluate the clinical utilization of skin Cholesterol (SC) for cardiovascular risk assessment in asymptomatic individuals at low, intermediate and high risk based on Framingham global risk estimates.

Preliminary studies have suggested that SC is an easy to measure, noninvasive marker of cardiovascular risk. This study is intended to provide further data in support of broader clearance by the Food and Drug Administration for the use of SC as a tool to identify asymptomatic patients at increased risk of cardiovascular disease. Currently, SC testing is cleared for use as part of risk assessment in subject suspected of having significant multi-vessel disease.

The current study data will be used to support the use of SC testing as part of cardiovascular risk assessment in subjects without suspected coronary artery disease (CAD).

DETAILED DESCRIPTION:
* The primary objective of the study will be to determine the relationship between skin cholesterol levels and carotid artery intima-media thickness (CIMT), a surrogate marker for atherosclerotic burden used as the "gold standard" comparator.
* Secondary objectives of the study will be to compare the skin cholesterol levels with other markers of CAD as HDL cholesterol, Apo B, hsCRP, and lipoprotein-association phospholipase A2.
* Another objective is to determine the relationship between skin cholesterol levels and the presence of carotid plaques detected by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent from the subject prior to testing.
* Males or females 30-80 years of age

Exclusion Criteria:

* 1. Known coronary heart disease, (history of myocardial infarction, coronary bypass surgery, coronary angioplasty, or angina pectoris with a positive stress test or angiographic documentation)
* Known peripheral vascular disease (claudication with ankle-brachial index < 0.9, angioplasty, or peripheral artery bypass procedure)
* Known cerebrovascular disease (stroke or TIA with documented carotid or aortic atherosclerosis)
* History of carotid artery endarterectomy or carotid artery surgery
* Diabetes mellitus (fasting glucose > 126 mg/dL, on on insulin-reducing medications)
* 10-year Framingham risk of cardiac death or MI using ATP III calculator >20%
* Subjects taking cholesterol-lowering medications
* Known hepatitis
* Known pregnancy
* Skin disease on either hand (e.g. eczema psoriasis, rash or broken skin)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary analysis will test if SC is a predictor of elevated CIMT (i.e. carotid wall thickness above the 75% percentile expected for subject's age sex and race based on projections from the Atherosclerosis Risk in Communities Study)

SECONDARY OUTCOMES:
Secondarily, estimates of relative risk will allow the comparison of the power of SC as a predictor and traditional risk and new emerging risk factors(hsCRP, Apo B100 and Phospholipase A2).

CONTACTS AND LOCATIONS:
Overall Officials: James H Stein, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States